CLINICAL TRIAL: NCT06897930
Title: A Phase 1b/2 Study of AZD0120, a Chimeric Antigen Receptor T-cell (CAR T) Therapy Targeting CD19 and B-cell Maturation Antigen (BCMA) in Subjects With Refractory Systemic Lupus Erythematosus (SLE)
Brief Title: A Study to Investigate the Safety, Tolerability, and Efficacy of AZD0120 in Adults With Refractory SLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8313C00001
Record Dates: First submitted 2025-03-12; First posted 2025-03-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: AZD0120; SLE; Systemic Lupus Erythematosus; Lupus; Lupus Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Drug: AZD0120 Single infusion of AZD0120
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD0120 (Experimental): Single dose of AZD0120
  Interventions: Biological: AZD0120; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: AZD0120 — Single infusion of AZD0120 on visit DAY 1 after completing required lymphodepleting chemotherapy..
  Other Names: GC012F
Drug: Cyclophosphamide — Lymphodepletion - specified dose prior to receiving AZD0120
Drug: Fludarabine — Lymphodepletion - specified dose prior to receiving AZD0120

SUMMARY:
This is a Phase 1b/2, single-arm, open-label, multi-center, clinical study of AZD0120, a CD19/BCMA dual CAR T cell therapy, to evaluate the safety, tolerability, and efficacy in adult participants with refractory Systemic Lupus Erythematosus.

DETAILED DESCRIPTION:
The study will enrol adult participants with refractory Systemic Lupus Erythematosus (SLE) The study will be run in 2 parts;

First part is Phase 1b during which the study aims to assess safety and tolerability of AZD0120 in patients in refractory SLE cohorts

Second part is Phase 2, during which the study aims to assess safety, tolerability and efficacy of the selected dose, following Phase 1b completion, in patients with refractory SLE

ELIGIBILITY:
INCLUSION:

1. Males or females aged 18 through 70 years inclusive at the time of consent.
2. Written informed consent in accordance with federal, local, and institutional guidelines.
3. Must be able and willing to adhere to the study visit schedule and other protocol requirements
4. Adequate hepatic, renal, pulmonary, and cardiac function
5. Have a clinical diagnosis of SLE according to the EULAR/ American College of Rheumatology (ACR) 2019 criteria with a positive ANA ≥1:80 and a score ≥10.
6. Have used at least two standard immunosuppressants (including one biological agent).
7. SLEDAI-2K score ≥6 at screening.
8. Must include a significant SLE related organ involvement: arthritis, myositis, rash, alopecia, mucosal ulcers, pleurisy, pericarditis, vasculitis, or renal.
9. For lupus nephritis: Diagnosis of proliferative lupus nephritis based on a renal biopsy obtained within 6 months prior to signing the informed consent form or during the screening period Class III, IV or V LN according to the WHO 2003 ISN/RPS classification.

EXCLUSION:

1. Have received prior treatment with CAR T therapy directed at any target.
2. Have received any therapy that is targeted to CD19 and/or BCMA
3. Received allogenic stem cell transplant or autologous stem cell transplant.
4. An active malignancy that is progressing or requires active treatment.
5. Primary immunodeficiency
6. Active viral or bacterial infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
PHASE 1B: To evaluate the safety and tolerability of AZD0120 in participants with refractory systemic lupus erythematosus (SLE) | 2 years
  The incidence and severity of adverse events (AEs)
PHASE 1B: Recommended Phase 2 Dose (RP2D) of AZD0120 in for Phase 2 | 2 years
  To determine the recommended phase 2 dose (RP2D) of AZD0120
PHASE 2: To evaluate the efficacy of AZD0120 in participants with refractory SLE | 2 years
  Proportion of participants achieving SRI-4 response

SECONDARY OUTCOMES:
PHASE 1B & 2: To evaluate the efficacy of AZD0120 in participants with refractory SLE | 2 years
  Proportion of participants achieving SLE Responder Index 4 (SRI-4) response over time
PHASE 1B & 2: To evaluate the efficacy of AZD0120 in participants with refractory SLE | 2 years
  Proportion of participants achieving remission in SLE (DORIS) remission over time
PHASE 1B & 2: To evaluate the efficacy of AZD0120 in participants with refractory SLE | 2 years
  Proportion of participants achieving Lupus Low Disease Activity State (LLDAS) over time
PHASE 1B & 2: To evaluate the efficacy of AZD0120 in participants with refractory SLE | 2 years
  Proportion of participants achieving British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) response over time
PHASE 1B & 2: To evaluate the efficacy of AZD0120 in participants with refractory SLE | 2 years
  Time from AZD0120 infusion and time from response to first disease flare
PHASE 1B & 2: To characterize the cellular kinetics of AZD0120 in participants with refractory SLE | 2 years
  The area under the concentration-time curve (AUC) from time zero (T0) to the last measurable concentration time point (AUClast)
PHASE 1B & 2: To characterize the cellular kinetics of AZD0120 in participants with refractory SLE | 2 years
  Area under the blood concentration-time curve from time zero to 28 days after dosing (AUC(0-28D))
PHASE 1B & 2: To characterize the cellular kinetics of AZD0120 in participants with refractory SLE | 2 years
  The last measurable concentration of AZD0120 (Clast)
PHASE 1B & 2: To characterize the cellular kinetics of AZD0120 in participants with refractory SLE | 2 years
  Maximum observed blood concentration (Cmax)
PHASE 1B & 2: To characterize the cellular kinetics of AZD0120 in participants with refractory SLE | 2 years
  Terminal half-life of a drug during its elimination phase in pharmacokinetics (t1/2λz)
PHASE 1B & 2: To characterize the cellular kinetics of AZD0120 in participants with refractory SLE | 2 years
  Time of the last measurable (quantifiable) concentration of a AZD0120 (Tlast)
PHASE 1B & 2: To characterize the cellular kinetics of AZD0120 in participants with refractory SLE | 2 years
  Time of maximum observed blood concentration (Tmax)
PHASE 1B & 2: To assess immunogenicity of AZD0120 | 2 years
  Presence of AZD0120 antibodies
PHASE 1B & 2: To determine whether replication-competent lentivirus is present in participants that receive AZD0120 | 2 years
  Presence of replication-competent lentivirus (RCL)
PHASE 2: To further characterize the safety of AZD0120 in participants with refractory SLE | 2 years
  Further characterization of the safety of AZD0120 by measuring the incidence and severity of Treatment Emergent Adverse Events (TEAEs)
PHASE 2: To assess changes from baseline for reported health-related quality of life, overall health status | 2 years
  To assess changes from baseline for Changes in Lupus Quality of life (LupusQoL)
PHASE 2: To assess changes from baseline for reported health-related quality of life, overall health status | 2 years
  To assess changes from baseline for FUNCTIONAL ASSESSMENT OF CHRONIC ILLNESS THERAPY (FACIT)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Darlinghurst
  - Research Site, Melbourne